CLINICAL TRIAL: NCT04573088
Title: Impact of Perioperative Acceptance-based Intervention on Early Psychological and Fanctional Recovery of Colorectal Cancer Patients
Brief Title: Acceptance-based Intervention at Colorectal Cancer Patients
Acronym: ABICOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, George Theodoropoulos, Associate Professor of Surgery, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB6/26-2-2019
Record Dates: First submitted 2020-09-16; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Colorectal Neoplasms; Acceptance Process; Pain, Procedural
MeSH Terms: conditions — Colorectal Neoplasms; Behavior; Pain, Procedural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABICOL (Experimental): 24 hours prior to surgery the patients undergo acceptance-based intervention, incorporating questions about their subjective perception about the surgery, the domains of their lives that have been affected, and on their own expectations from surgery and its effects on their lives. They will be asked to express their fears and worries about their condition and they will be discussed about the likelihood of experiencing postoperative pain.
  Interventions: Behavioral: ACCEPTANCE-BASED INTERVENTION
- CONTROL (No Intervention): No acceptance-based intervention or other discussion related to the patients' fears and worries will be applied.

INTERVENTIONS:
Behavioral: ACCEPTANCE-BASED INTERVENTION — 24 hours prior to surgery the patients undergo acceptance-based intervention, incorporating questions about their subjective perception about the surgery, the domains of their lives that have been affected, and on their own expectations from surgery and its effects on their lives. They will be asked to express their fears and worries about their condition and they will be discussed about the likelihood of experiencing postoperative pain.
  Arms: ABICOL

SUMMARY:
Taking into account the unavoidable effect of a major oncologic surgery commonly required for colorectal cancer patients and the recognized psychological and functional sequelae of the surgical treatment on their status, we will evaluate the influence of a psychological intervention, known as acceptance-based intervention, offered to those patients at the preoperative setting. Reduction of anxiety and assessmemt of indices of post-intervention psychological and functional recovery will be the primary goals of the study.

DETAILED DESCRIPTION:
Introduction: Uncertainty, fears and anxiety are common reactions to an upcoming colectomy for colorectal cancer patients and are related not only to cancer disease, but also to the inevitable change in colon anatomy, affecting their preoperative psychological and functional condition and their postsurgical recovery.

Purpose: We aim to evaluate the psychological and functional recovery of colorectal cancer patients, who undergo colectomy, after an acceptance-based nursing intervention. The scope of this brief preoperative intervention is to enable patients to cope more efficiently with the upcoming surgery and their health status, as it is expected to reduce anxiety and have positive effect on postsurgical psychological and functional recovery.

Methods: The study includes histologically diagnosed patients with colorectal cancer, regardless of stage, who are scheduled to undergo colectomy. Patients will be divided into two groups-the experimental and the control group-by simple randomization. Both groups are going to complete a set of same questionnaires regarding quality of life, sleep, anxiety, depression and functional status. Patients in the control arm will then receive treatment-as-usual while patients in the experimental arm will also receive an acceptance-based intervention before surgery. Postoperatively, for both groups, apart from the self-reported symptoms, we will assess objective recovery factors, such as postoperative complications

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven colorectal adenocarcinoma
* Age > 18 years

Exclusion Criteria:

* Metastasis at time of diagnosis
* Recurrence at time of diagnosis
* History of other malignancies
* Mental retardation
* Deafness
* Illiteracy
* ASA score>3
* Poor performance status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-06-22 (Estimated); Study Completion 2022-01-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain as measured by VAS score | Third postoperative day
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations.The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured orientated from the left (worst) to the right (best).

SECONDARY OUTCOMES:
Functional status as measured by "Maintain Function" Scale (MFS) | Third postoperative day
  "Maintain function" scale is a validated 5-item summative. Each item begins with the stem, "How confidant are you that you know or can," and assesses an aspect of daily life-function, such as work and social activities. The responses are a 5-level Likert scale from 0 = "not at all confident" to 4 = "completely confident." We did not include a "not applicable" response option. The self-efficacy scores range between 0 and 20, with a higher score indicating better self-efficacy to maintain function.
Anxiety and depression measured by Brief Illness Perception Questionnaire (Brief IPQ) | Third postoperative day
  The Brief Illness Perception Questionnaire (Brief IPQ) is a 9-item questionnaire designed to rapidly assess cognitive and emotional representations of illness. The Brief IPQ uses a single-item scale approach to assess perception on a 0-10 response scale. The Brief IBQ comprises 5 items on cognitive representation of illness perception: consequences, timeline, personal control, treatment control, and identity. There are 2 items on emotional representation: concern and emotions. One item is on illness comprehensibility. The last item is on perceived cause of illness, in which respondents list the three most important causal factors in their illness.
Anxiety and depression measured by State-Trait Anxiety (STAI) questionnaire | Third postoperative day
  The State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic. Higher scores are positively correlated with higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: George E Theodoropoulos, Principal Investigator — Associate Professor of Surgery
Locations (1):
- NKUAthens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes
Sharing clinical trial data with other professional organizations and researchers will be important element to support best practice principles in our clinical trial.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At completion of study and analysis of results
Access Criteria: If requested for universal prospective registration If requested by journals for publication If requested by researchers running similar clinical trials